CLINICAL TRIAL: NCT03194100
Title: Comparison of Serum METRNL Concentration Between Type 2 Diabetes and Normal Glucose Tolerance
Brief Title: Serum METRNL Concentration in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Bon Jeong Ku, Professor, Chungnam National University Hospital
Other Study IDs: METRNL
Record Dates: First submitted 2017-06-18; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetes Mellitus
- Prediabetes
- Normal glucose tolerance

SUMMARY:
The investigators measured serum METRNL levels in newly diagnosed patients with type 2 diabetes (T2DM) compared with normal glucose tolerance or prediabetes and explored the correlations between its serum levels and various metabolic parameters

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have not been diagnosed diabetes mellitus

Exclusion Criteria:

* Person with diabetes who were treated with oral hypoglycemic agent or insulin
* Individuals with type 1 diabetes, gestational diabetes, active hepatitis/liver cirrhosis, chronic renal failure on hemodialysis, congestive heart failure, or other known major disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Oral glucose tolerance test (OGTT) was performed in all of the included participants. The participants were divided into three groups according to the American Diabetes Association criteria; normal glucose tolerance, prediabetes and diabetes mellitus.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
serum METRNL concentration | on the 1 day of oral glucose tolerance test